CLINICAL TRIAL: NCT07279805
Title: Peripheral Perfusion Index as a Predictor of Post-spinal Hypotension in Patients Undergoing Lower Limb Surgeries
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: fmasu ms579/2024
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-08

CONDITIONS: Post Spinal Anaesthesia Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study was carried out on a sample of 40 patients over a period of 6 months to asses the peripheral perfusion index as a Predictor for post spinal hypotension in patient undergoing lower limp surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aging between 21-40 years of both sexes with average weight of 60-80 kg, and average height of 160-180.

  * Patients undergoing Elective Lower limb Surgeries under successful spinal anesthesia (duration of surgery 45-120 minutes).
  * ASA physical status classes I - II.

Exclusion Criteria:

* Patient's refusal of procedure or participation in the study.

  * ASA classes III or above. Coagulopathy and bleeding disorders.
  * Body mass index >40kg/m2
  * Contraindications to spinal anesthesia.
  * Hypersensitivity to the study medications.
  * Patients receiving vasoactive drugs.
  * Patients undergoing emergency surgery.
  * Duration more than 2hours.
  * Major bleeding.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients undergoing elective lower limb surgeries at El-demerdash Hospital of Surgery during the study period. Surgeries include Anterior/Posterior curciate ligament repair,knee arthroscopy,Hip and Knee replacement,tendon repair and varicose veins ligation.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2025-03-09 (Actual)

PRIMARY OUTCOMES:
Assess the ability of baseline peripheral perfusion index to predict post spinal hypotension spinal anesthesia-induced hypotension in patients undergoing lower limb surgeries | during the operation time.
  Assess the ability of baseline peripheral perfusion index to predict post spinal hypotension

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams University, Cairo, Egypt